CLINICAL TRIAL: NCT00371098
Title: Prospective, Randomized, Double-Blind Placebo Controlled Study on Influenza Vaccination in Prevention From Coronary Events in Patients With Coronary Artery Disease Confirmed by Angiography
Brief Title: Influenza Vaccination in Prevention From Acute Coronary Events in Coronary Artery Disease - FLUCAD Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Collaborators: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IK-NP-0021-2/812/04; 2 P05B 016 27
Record Dates: First submitted 2006-08-31; First posted 2006-09-01 (Estimated); Last update posted 2007-10-23 (Estimated); Status verified 2007-10

CONDITIONS: Coronary Artery Disease
Keywords: influenza vaccination; coronary artery disease; prevention; acute coronary syndromes
MeSH Terms: conditions — Coronary Artery Disease; Influenza, Human; Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active vaccine (Experimental): patients received active influenza vaccine for season 2004/2005
  Interventions: Biological: Influenza vaccination: Influvac (SolvayPharma)
- placebo vaccine (Placebo Comparator): patients received placebo influenza vaccine for season 2004/2005 containing all vaccine compounds except viral antigens
  Interventions: Biological: placebo influenza vaccine

INTERVENTIONS:
Biological: Influenza vaccination: Influvac (SolvayPharma)
  Arms: active vaccine
Biological: placebo influenza vaccine
  Arms: placebo vaccine

SUMMARY:
Background: Influenza vaccination is recommended in patients (pts) with cardiovascular disease, however there is a shortage of clinical studies proving its protective effect on clinical course of coronary artery disease (CAD). The aim of the study was to evaluate the effect of influenza vaccination on the incidence of coronary events in pts with CAD confirmed by coronary angiography.

DETAILED DESCRIPTION:
A possible relation between influenza and higher mortality from cardiovascular problems was first noticed in early nineteen hundreds, after epidemics in Europe and United States were discovered (1). In the last decade many studies implicating an important role of inflammation and infection (Herpes virus, Chlamydia pneumoniae, Helicobacter pylori) in development and progression of atherosclerosis (2,3), and markers of inflammation like: hs-CRP, fibrinogen, have become new independent cardiovascular risk factors (4).

Many general physicians now recommend influenza vaccination in patients with coronary artery disease (CAD) despite shortage of studies proving its protective effect on clinical course of CAD. In literature we found only a few reports exploring the hypothesis that influenza vaccination might reduce the incidence of myocardial infarction (MI) and acute coronary syndromes (ACS).

Naghavi et all. in retrospective, case- control study of 218 patients with chronic coronary disease reported that influenza vaccination was strongly associated with freedom from new MI during the same influenza season. (OR 0.33, 95% CI 0.13 to0.82, p=0.017) (5). Gurfinkiel et all. evaluated in prospective, single- blind Fluvacs study that preventive impact of vaccination on subsequent ischemic events at 6 months follow-up. Study group consisted of 301 patients after coronary angioplasty (PCI). The first primary outcome- cardiovascular death occurred in 2% in vaccine group compared with 8% in the control group (p=0.01) and triple composite end point (death, myocardial infarction and hospitalization from ischemia occurred in 11% in vaccine group vs. 23% in controls (p=0.0009) (6). In the contrary, Jackson et all. in largest study of 1378 survivors of first MI, in long (median 2.3 year) follow-up didn't find the benefit of influenza vaccine on the protection against recurrent coronary events (7).

The aim of our study is to evaluate the influence of influenza vaccination on the incidence of cardiac events (cardiovascular death, myocardial infarction, acute coronary syndromes, coronary revascularization and hospitalizations from ischemia) in patients with angiographically confirmed coronary disease.

References:

1. Collins SD. Excess mortality from causes other that influenza and pneumonia during influenza epidemics. Public Health Rep. 1932;47:2159-80.
2. Sorlie PD, Adam E, Melnick SL, et al. Cytomegalovirus/herpesvirus and carotid atherosclerosis: the ARIC Study. J Med Virol. 1994;42:33-37.
3. Zhou YF, Wanishsawad C, Epstein SE. Chlamydia pneumonia-induced transaction of cytomegalovirus: potential synergy of infectious agents in the pathogenesis of atherosclerosis. J Am Coll Cardiol. 1999;33(suppl A):260A.
4. Toss H, Lindahl B, Siegbahn A, Wallentin L. (Frisc study group). Prognostic Influence of Increased Fibrinogen and C- reactive Protein Levels in Unstable Coronary Artery Disease. Circulation 1997; 96: 4304- 4210.
5. Naghavi M., Barlas Z., Siadaty S., Nagiub S., Madjid M., Casscells W.: Association of influenza vaccination and reduced risk of myocardial infarction Circulation 2000; 102:3039-3045.
6. Gurfinkel E.P., Leon de la Fuente R., Mendiz O., Mautner B. For the FLUVACS Study Group: Influenza vaccine pilot study in acute coronary syndromes and planned percutaneous coronary interventions. The FLU vaccination acute coronary syndromes (FLUVACS) Study. Circulation 2002;105:2143-2147.
7. Jackson L.A., Heckbert S.R., Psaty B.M., Malais D., Barlow W.E., Thompson W.W. Vaccine Safety Datalink Study Group: Influenza vaccination is not associated with a reduction in the risk of recurrent coronary events. Am. J. Epidemiol. 2002; 156: 634-40.

ELIGIBILITY:
Inclusion Criteria:

* Patients, aged 30-80 years, with CAD confirmed by coronarography with at least 50% stenosis of one large epicardial coronary artery.

Exclusion Criteria:

* planned cardiovascular surgery within 6 months, congestive heart failure NYHA III/IV, evolving renal failure, neoplastic disease, psycho-organic disorder or any factor impeding follow-up, contraindication to vaccination.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 658 (Actual)
Dates: Start 2004-10; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
cardiovascular death | 12 months

SECONDARY OUTCOMES:
First composite study end point was Major Adverse Cardiac Event (MACE). MACE was combined of: cardiovascular death, acute myocardial infarction (MI), coronary revascularization (PCI or coronary bypass). | 12 month
Second composite study end point was Ischemic Event (MACE or hospitalization for ischemia). | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Ciszewski, MD, PhD, Principal Investigator — 1st Dept of Coronary Artery Disease, Institute of Cardiology, Warsaw, Poland
Locations (1):
- 1st Dept. of Coronary Artery Disease, Institute of Cardiology, Warsaw, Poland

REFERENCES:
- [Result] Ciszewski A, Bilinska ZT, Brydak LB, Kepka C, Kruk M, Romanowska M, Ksiezycka E, Przyluski J, Piotrowski W, Maczynska R, Ruzyllo W. Influenza vaccination in secondary prevention from coronary ischaemic events in coronary artery disease: FLUCAD study. Eur Heart J. 2008 Jun;29(11):1350-8. doi: 10.1093/eurheartj/ehm581. Epub 2008 Jan 10. PMID 18187561
- See also: Institute of Cardiology, Warsaw, Poland — http://www.ikard.pl